CLINICAL TRIAL: NCT03067922
Title: Post Mastectomy Pain Syndrome at an Indian Tertiary Cancer Centre: Incidence, Pain Severity, Impact on Daily Function and Quality of Life
Brief Title: Postmastectomy Pain Syndrome in an Indian Cancer Hospital
Status: Completed | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Aparna Chatterjee, Professor, Tata Memorial Centre
Other Study IDs: TataMC
Record Dates: First submitted 2017-02-10; First posted 2017-03-01 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Pain Syndrome; Mastectomy; Quality of Life
Keywords: Mastectomy; Pain; Severity; Life quality
MeSH Terms: conditions — Somatoform Disorders; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non interventional study — Not applicable. No intervention will be done. it is an observational study assessing pain after mastectomy and the quality of life as assessed from validated questionnaires given to the patients at regular intervals

SUMMARY:
Breast cancer is the most common cancer in women in India and accounts for 27% of all cancers in women. Incidence rises in early thirties, peaks at 50-64 years. Approximately 48% are below 50 years of age. Most present when symptoms develop, so are 2B and beyond. Treatment depends on the stage of the disease. Surgical removal of the tumour is part of the treatment attempting a cure.

Simple mastectomy involves removal of breast tissue without axillary lymph node dissection or removal of chest wall muscles. Radical mastectomy involves removal of the entire breast, skin, pectoralis major and minor muscles and ipsilateral axillary lymph nodes. Modified radical mastectomy involves removal of the breast and ipsilateral axillary lymph nodes. The pectoralis muscle is preserved. Breast conserving surgery involves removal of tumour with or without axillary dissection. The extent of surgery tells us about the nerve damage, local tissue handling. For example operating in upper and outer quadrant of breast and axilla increases nerve handling in that particular region. Local radiation also plays a role.

Persistent pain after mastectomy was first reported in the 1970s by Wood and defined by International Association for Study of Pain (IASP) as pain in the anterior aspect of the thorax, axilla, and/or upper half of the arm beginning after mastectomy or quadrantectomy and persisting for more than three months after surgery and known as Postmastectomy pain Syndrome (PMPS). It is a common problem, with a 25- 60% incidence. The pain is described as burning or tenderness with paroxysms of lancinating, shock-like pain, and also described by some as dysesthesia (perception of non noxious stimuli as painful). Risk factors for PMPS include age, raised Body mass index (BMI), severity of postoperative pain, type of surgery, susceptibility to pain with a history of other pains such as headache and dysmenorrhoea. Axillary hematoma and postoperative radiotherapy have also been implicated in the development of PMPS.

Tata Memorial Hospital, is a tertiary cancer institute in India. Around 4000 patients with suspected breast cancers register annually at the hospital and approximately 2800 breast cancer surgeries are performed yearly. Very few studies on PMPS in Indian population exist. We therefore plan to identify the incidence of PMPS in our patients and also the severity of pain along with its impact on daily function and quality of life

DETAILED DESCRIPTION:
Tata Memorial Hospital, a 629 bed tertiary cancer institute conducts approximately 6000 surgeries per year. Approximately 4000 (4239 in 2015) patients with suspected breast cancers register annually at the hospital and around 2800 breast cancer surgeries are performed every year. Very few studies on PMPS in Indian population exist. The investigators therefore, aim to identify the incidence of post mastectomy pain syndrome PMPS) in this population. The investigators also aim to identify the severity of postmastectomy pain along with its impact on daily function and quality of life.

STUDY DESIGN:

Prospective study over 12 months with follow up until 6th month from enrollment with interim analysis in the month of November for presentation of the CoPI's thesis.

MATERIALS & METHODS:

Prospective study over a period of 12 months from commencement of study after Institutional ethics committee approval, at Tata Memorial hospital and ACTREC. Female patients scheduled for undergoing surgery for breast cancer conservative and radical and willing to participate will be enrolled in the study after obtaining a written informed consent. Pain scores will be assessed using Numerical rating scale [with pain score 1-3 mild, 4 to 6 moderate and 7 and above severe]. History of predisposition to recurrent headaches and dysmenorrhea will be noted. Details of disease stage, chemotherapy and/or radiotherapy will also be documented from the Electronic medical records. Analgesia will be managed by the primary surgical team as is currently being done. The analgesia administered to the patient will also be recorded. participants noted to have moderate to severe pain despite analgesics prescribed by the surgical team will be referred to the acute pain service (APS) for further management.

Postoperative pain severity both the average & worst pain will be recorded at discharge from hospital, 1st, 4th and 6th month after the surgery. The Details of postoperative pain analgesic use and effect on daily function will be documented with the help of postal cards with questionaires in envelop addressed to the investigators. Study will emphasize on the type, severity, the site of pain whether, lateral or anterior chest wall, axilla, ipsilateral medial upper arm or back, the type of pain (burning, tingling, shooting, stabbing etc) and effects on daily function and quality of life. Details of postoperative hematoma, infection, local recurrence will also be recorded from the history, electronic medical records and documents of participants. Details of postoperative chemotherapy and radiation will also be obtained from patient's notes and the electronic medical record All participants will be administered the short form of the Brief Pain inventory [BPI], EORTC QLQ 30, preoperatively, at 1 month, 4 months & 6 months after surgery.

The Brief pain inventory {BPI} (obtained with permission from MD Anderson), which assesses the severity of pain and impact of pain on daily functions will be administered to the participant in the language familiar to them, preoperatively, at 1 month, 4th and 6th month postoperatively. The short form comprises of nine questions related to the severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week.It has been widely used and validated in several languages the world over.

EORTC QLQ [Quality of life Questionaries ] is an integrated system for assessing quality of life [health related ]. This self administered questionnaires incorporates five functional scales, physical [PF], role [RF], cognitive [CF], emotional [ef], and social; three symptoms scale for fatigue, pain and nausea/vomiting; a global health quality of life scale and several single items for financial impact and additional symptoms like diarrhea, appetite loss, sleep disturbance. This would help identify the quality of life of the participants and its affection.

If a participant cannot follow up at the said intervals, the pain scores would be obtained telephonically and the BPI, EORTC QLQ 30 form in prepaid envelopes would be given to them at discharge which they would have to duly fill in and post them to the given address at the appropriate intervals. If the next follow up to the hospital coincides with the 4th or 6th postoperative month, the participant will visit the pain clinic for an assessment and completing the BPI.

ELIGIBILITY:
Inclusion Criteria:

* Female patient undergoing mastectomy simple radical with or without axilla dissection
* Literate and can read and write in either English, Hindi, Marathi
* Willing to fill forms and post them and/or answer questions on phone

Exclusion Criteria:

* Refusal of consent
* Patient who has previously undergone major surgery around breast and chest wall
* Benign breast pathology
* Patient's with impaired cognitive function
* Emergency surgery
* PECs block study (PECTORALIS BLOCK)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients scheduled for undergoing surgery for breast cancer conservative and radical and willing to participate will be enrolled in the study after obtaining a written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Post mastectomy pain syndrome (PMPS) | 6 months after surgery
  presence of pain around the mastectomy site and ipsilateral arm after the mastectomy

SECONDARY OUTCOMES:
pain severity | At 1 month after surgery
  How severe the pain is after mastectomy from the Pain intensity obtained from the Brief Pain inventory questionnaire
pain severity | At 4 months after surgery
  How severe the pain is after mastectomy from the pain intensity obtained from the Brief Pain inventory questionnaire
pain severity | At 6 months after surgery
  How severe the pain is after mastectomy from the pain intensity obtained from the Brief Pain inventory questionnaire
Impact on daily function | At 1 month after surgery
  How the pain after mastectomy per se affects day to day functioning of the patient and how the quality of her life is affected. The impact of pain on daily life will be identified from the Brief Pain inventory questionnaire which the patient would have to complete at this time point.
Impact on quality of life | At 1 month after surgery
  The impact of the mastectomy on Quality of life of the patient would be assessed from the EORTC-QLQ 30 questionnaire completed by the patient
Impact on daily function | At 4 months after surgery
  How the pain per se affects day to day functioning of the patient.The impact of pain on daily life will be identified from the Brief Pain inventory questionnaire which the patient would have to complete at this time point.
Impact on quality of life | At 4 months after surgery
  The impact of the mastectomy on the quality of life of the patient would be assessed from the EORTC-QLQ 30 questionnaire completed by the patient at his time point.
Impact on daily function | At 6 months after surgery
  How the pain per se affects day to day functioning of the patient .The impact of pain on daily life will be identified from the Brief Pain inventory questionnaire which the patient would have to complete at this time point.
Impact on quality of life | At 6 months after surgery
  the impact of teh mastectomy on the quality of life of the patient would be assessed from the EORTC-QLQ 30 questionnaire completed by the patient at this time point.

CONTACTS AND LOCATIONS:
Overall Officials: APARNA S CHATTERJEE, MD,FCARCSI, Principal Investigator — Tata Memorial Centre
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith WC, Bourne D, Squair J, Phillips DO, Chambers WA. A retrospective cohort study of post mastectomy pain syndrome. Pain. 1999 Oct;83(1):91-5. doi: 10.1016/s0304-3959(99)00076-7. PMID 10506676
- [Result] Couceiro TC, Menezes TC, Valenca MM. Post-mastectomy pain syndrome: the magnitude of the problem. Rev Bras Anestesiol. 2009 May-Jun;59(3):358-65. doi: 10.1590/s0034-70942009000300012. English, Portuguese. PMID 19488550
- [Result] Mejdahl MK, Andersen KG, Gartner R, Kroman N, Kehlet H. Persistent pain and sensory disturbances after treatment for breast cancer: six year nationwide follow-up study. BMJ. 2013 Apr 11;346:f1865. doi: 10.1136/bmj.f1865. PMID 23580693
- [Result] Bray F, Ren JS, Masuyer E, Ferlay J. Global estimates of cancer prevalence for 27 sites in the adult population in 2008. Int J Cancer. 2013 Mar 1;132(5):1133-45. doi: 10.1002/ijc.27711. Epub 2012 Jul 26. PMID 22752881
- [Result] Wood KM. Intercostobrachial nerve entrapment syndrome. South Med J. 1978 Jun;71(6):662-3. doi: 10.1097/00007611-197806000-00016. PMID 663696
- [Result] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Result] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Result] Miguel R, Kuhn AM, Shons AR, Dyches P, Ebert MD, Peltz ES, Nguyen K, Cox CE. The effect of sentinel node selective axillary lymphadenectomy on the incidence of postmastectomy pain syndrome. Cancer Control. 2001 Sep-Oct;8(5):427-30. doi: 10.1177/107327480100800506. PMID 11579339
- [Result] Steegers MA, Wolters B, Evers AW, Strobbe L, Wilder-Smith OH. Effect of axillary lymph node dissection on prevalence and intensity of chronic and phantom pain after breast cancer surgery. J Pain. 2008 Sep;9(9):813-22. doi: 10.1016/j.jpain.2008.04.001. Epub 2008 Jun 30. PMID 18585963
- [Result] Glechner A, Wockel A, Gartlehner G, Thaler K, Strobelberger M, Griebler U, Kreienberg R. Sentinel lymph node dissection only versus complete axillary lymph node dissection in early invasive breast cancer: a systematic review and meta-analysis. Eur J Cancer. 2013 Mar;49(4):812-25. doi: 10.1016/j.ejca.2012.09.010. Epub 2012 Oct 17. PMID 23084155